CLINICAL TRIAL: NCT07224594
Title: Comparing Optimized Models of Primary And Specialist Services for Palliative Care
Acronym: COMPASS-PC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Principal Investigator, Scott Halpern, John M. Eisenberg Professor of Medicine, Epidemiology, and Medical Ethics & Health Policy, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 855378; PLACER-2022C3-30553 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2025-10-24; First posted 2025-11-04 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Seriously Ill Hospitalized Patients
Keywords: Palliative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standardized Usual Care (Active Comparator): Active control group, where high-risk patients (i.e., with a 1-year mortality risk between 70% and 94%) will receive usual care. A specialist PC consult is ordered by default for the very high-risk patients (i.e., 1-year mortality risk ≥ 95%), unless clinicians cancel the order.
  Interventions: Behavioral: Standardized Usual Care
- Trained Generalist Palliative Care (Experimental): Generalist clinicians trained in PC domains receive an EHR-based alert to document whether or not they have addressed PC domains for high-risk patients ('accountable justification intervention'). A specialist PC consult is ordered by default for the very high risk patients (i.e., 1-year mortality risk ≥ 95%) unless clinicians cancel the order.
  Interventions: Behavioral: Default Order; Behavioral: Accountable Justification
- Specialist Palliative Care (Experimental): A specialist PC consult is ordered by default for all patients with a ≥ 70% 1-year mortality risk ('default order intervention'), unless clinicians cancel the order.
  Interventions: Behavioral: Default Order

INTERVENTIONS:
Behavioral: Default Order — A specialist PC consult is automatically ordered for patients meeting a certain threshold of 1-year mortality risk (dependent on arm). An EHR-based Our Practice Advisory (OPA) alert on Open Chart informs clinicians when the default order will become active, and how to cancel an order within 24 hours if they elect to do so.
  Arms: Specialist Palliative Care; Trained Generalist Palliative Care
Behavioral: Accountable Justification — An EHR-based Our Practice Advisory alert asks generalist clinicians to self-report whether they have provided primary PC by clicking which of 4 key PC domains they have addressed or to provide a brief justification as to why not.
  Arms: Trained Generalist Palliative Care
Behavioral: Standardized Usual Care — High-risk patients (i.e., with a 1-year mortality risk between 70% and 94%) will receive usual care. For very high-risk patients (i.e., with a 1-year mortality risk of ≥ 95%), an EHR-based Our Practice Advisory (OPA) alert on Open Chart informs clinicians when the default order will become active, and how to cancel an order within 24 hours if they elect to do so.
  Arms: Standardized Usual Care

SUMMARY:
Palliative care (PC) seeks to reduce suffering and improve quality of life for patients with serious illnesses and their families. National guidelines recommend that clinicians either provide palliative care themselves (generalist PC) or consult experts (specialist PC) as a standard part of serious illness care. This pragmatic clinical trial will be conducted with 48 hospitals at two large U.S. health systems and enroll more than 78,000 seriously ill hospitalized patients. Eligibility is determined by a mortality prediction score where enrolled patients have at least a 70% risk of dying within 1 year. Enrollment assessment occurs as close as possible to 36 hours post admission. The 48 hospitals will be randomized to 3 arms: (1) standardized usual care, (2) trained generalist PC, or (3) specialist PC. Generalist clinicians are trained using the Center to Advance Palliative Care (CAPC) online trainings. This pragmatic, hybrid effectiveness-implementation parallel-cluster RCT will assess the comparative effectiveness of triggering generalist PC and specialist PC on several patient-centered outcome measures, and follows a pilot feasibility study. We will collect Patient-Reported Outcomes (PROs) surveys from a random subset of enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older; AND Predicted 1-year mortality risk of 70% or greater; AND Admitted to a study hospital.

Exclusion Criteria:

* Patients who die or have an active or completed discharge order prior to enrollment time OR
* Readmission within 182 days of an eligible encounter OR
* Ineligible service line, with current admission status labeled as: hospice, acute rehabilitation, skilled nursing facility, long-term acute care, psychiatry, obstetrics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78302 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-11-01 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Hospital free days | Enrollment- 182 days.
  Count of days from enrollment spent alive outside of an acute care hospital through 182 days.

SECONDARY OUTCOMES:
Patient quality of life | 1-month, 3-months, and 6-months post-enrollment
  Patient or caregiver report of the patient's quality of life using the 15-item McGill Quality of Life survey instrument.
Clinician communication | 1-month post-enrollment
  Patient or caregiver report of how much patients feel heard and understood, using the 4-item CMS-MACRA survey instrument
Pain management | 1-month post-enrollment
  Patient or caregiver report of whether patients receive desired help for pain, using the 3-item CMS-MACRA survey instrument.
Goal concordant care | 1-month post-enrollment
  Patient or caregiver report of the patient's perception of whether their treatment matched what they wanted.
Social interaction | 1-month post-enrollment
  Patient or caregiver report of patient's social support using the 4-item Duke Social Support Index's Social Interaction Sub-scale
Loneliness | 1-month post-enrollment
  Patient or caregiver report of patient's loneliness using the 3-item Duke UCLA loneliness scale.
Hospital free days at 3 months | Enrollment - 3-months post-enrollment
  Count of days from enrollment spent alive and not in an acute care hospital through 3 months.
Institution free days at 3 months | Enrollment - 3-months post-enrollment
  Count of days from enrollment spent alive and not in any care facility through 3 months.
Institution free days at 6 months | Enrollment - 6-months post-enrollment
  Count of days from enrollment spent alive and not in any care facility through 6 months.
30-day hospital readmissions | Enrollment - 30 days post-enrollment
  Count of readmissions
90-day hospital readmissions | Enrollment - 90 days post-enrollment
  Count of readmissions.
Community-based palliative care use | Enrollment - 6-months post-enrollment
  Binary variable indicating any use (use/no use) captured through EHR and claims data and count of days of PC visits.
Hospice use | Enrollment - 6-months post-enrollment
  Binary variable indicating any use (use/no use) captured through EHR and claims data and count of days of hospice.
Change in code status | Enrollment- Discharge from hospital (an average of 7 days)
  Binary indicator of whether code status changed from enrollment.
Time to palliative care consult | Enrollment- Discharge from hospital (an average of 7 days)
  Time from enrollment until receipt of the first documented inpatient palliative care consultation note.

OTHER OUTCOMES:
End-of-Life Care | 3 months post-patient death
  Caregiver report of the patient's end-of-life experience using the 14-item Family Assessment of Treatment at the End of Life Short Form (FATE-S) survey instrument and two additional questions regarding place of death and whether it was their preferred location.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Halpern, MD, PhD, Principal Investigator — University of Pennsylvania; Katherine Courtright, MD, MS, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Kaiser Permanente Southern California, Pasadena, California
  - Trinity Health, Livonia, Michigan

IPD SHARING:
Plan to Share IPD: Yes
De-identified data (the Analyzable Data Set, Full Protocol, metadata, data dictionary, full statistical analysis plan (including all amendments and all documentation for additional work processes)), and analytic code from a PCORI-funded research project from this PCORI-funded clinical trial will be made available on the Patient-Centered Outcomes Data Repository.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The IPD and supporting information will be available between 3 and 6 months after the study completion date, and will be available on the Patient Centered Outcomes Data Repository in line with PCORI's policies for data retention.
Access Criteria: Applicants will follow the guidelines as set out on the Patient Centered Outcomes Data Repository for accessing this data set.
URL: https://www.pcori.org/research-related-projects/about-our-research/data-sharing-maximizing-utility-pcori-funded-data